CLINICAL TRIAL: NCT00895622
Title: Phase II Trial of Observation for Low-Risk Meningiomas and of Radiotherapy for Intermediate- and High-Risk Meningiomas
Brief Title: Observation or Radiation Therapy in Treating Patients With Grade I, Grade II, or Grade III Meningioma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Radiation Therapy Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH); NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RTOG-0539; CDR0000641815
Record Dates: First submitted 2009-05-07; First posted 2009-05-08 (Estimated); Results first posted 2018-01-19 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-08

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: adult grade I meningioma; adult grade II meningioma; adult grade III meningioma; adult anaplastic meningioma; adult papillary meningioma; recurrent adult brain tumor
MeSH Terms: conditions — Central Nervous System Neoplasms; Meningioma; Brain Neoplasms | interventions — Radiotherapy; Proton Therapy; Radiotherapy, Conformal; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Low Risk (No Intervention): No treatment given.
- Intermediate Risk (Experimental): 54 Gy radiotherapy
  Interventions: Radiation: 54 Gy radiotherapy
- High Risk (Experimental): 60 Gy radiotherapy
  Interventions: Radiation: 60 Gy radiotherapy

INTERVENTIONS:
Radiation: 54 Gy radiotherapy — External beam radiation therapy (EBRT) to a total dose of 54 Gy (RBE) in 30 fractions. 1.8 Gy (RBE) daily, 5 fractions per week, excluding weekends. 3D-CRT or IMRT or Proton allowed.
  Other Names: external beam radiation therapy (EBRT); radiation therapy (RT); Proton therapy; Three-dimensional conformal radiotherapy (3D-CRT); Intensity-modulated radiation therapy (IMRT)
  Arms: Intermediate Risk
Radiation: 60 Gy radiotherapy — External beam radiation therapy using intensity-modulated radiation therapy (IMRT) to a total dose of 60 Gy in 30 fractions. 2.0 Gy daily, 5 fractions per week, excluding weekends.
  Other Names: external beam radiation therapy (EBRT); radiation therapy; Intensity-modulated radiation therapy (IMRT)
  Arms: High Risk

SUMMARY:
RATIONALE: Sometimes a tumor may not need treatment until it progresses. In this case, observation may be sufficient. Specialized radiation therapy that delivers a high dose of radiation directly to the tumor, such as 3-dimensional conformal radiation therapy and intensity-modulated radiation therapy, may kill more tumor cells and cause less damage to normal tissue. It is not yet known whether observation is more effective than radiation therapy in treating patients with meningioma.

PURPOSE: This phase II trial is studying observation to see how well it works compared with radiation therapy in treating patients with grade I, grade II, or grade III meningioma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To estimate the rates of progression-free survival at 3 years in patients with low-risk meningioma undergoing observation and in patients with intermediate- or high-risk meningioma undergoing radiotherapy.

Secondary

* To study the concordance, or lack thereof, between central and parent institution histopathologic diagnosis, grading, and subtyping.
* To estimate the rates of overall survival at 3 years in these patients.
* To estimate the incidence rates of acute and late adverse events ≥ grade 2 in patients with intermediate- or high-risk meningioma undergoing radiotherapy.
* To evaluate MRI imaging predictors by central neuroradiology review at diagnosis, at any failure, and at 3 years.
* To evaluate adherence to protocol-specific target and normal tissue radiotherapy parameters.

This is a multicenter study. Patients are assigned to 1 of 3 groups according to risk.

After completion of study treatment, patients are followed up every 3-6 months for 3 years and then annually for 10 years.

ELIGIBILITY:
Inclusion Criteria:

1. A histologically documented World Health Organization (WHO) grade I, II, or III meningioma, newly diagnosed or recurrent, and of any resection extent, confirmed by central pathology review. Patients are partitioned according to three groupings: Group I (low risk), Group II (intermediate risk), and Group III (high risk) as defined below:

   * Group I (low risk): Patients with a newly diagnosed WHO grade I meningioma that has been gross totally resected (Simpson's grade I, II, or III resections, with no residual nodular enhancement on postoperative imaging) or subtotally resected (residual nodular enhancement or Simpson grade IV or V excision). The extent of resection will be based upon the neurosurgeons' assessment and postoperative MR imaging.
   * Group II (intermediate risk): Patients with a newly diagnosed gross totally resected WHO grade II meningioma or patients with a recurrent WHO grade I meningioma irrespective of the resection extent. Resection extent will be recorded on the same basis described above for the low-risk group.
   * Group III (high risk): Patients with a newly diagnosed or a recurrent WHO grade III meningioma of any resection extent; patients with a recurrent WHO grade II meningioma of any resection extent; or patients with a newly diagnosed subtotally resected WHO grade II meningioma. In the setting of a newly diagnosed meningioma, the histologic diagnosis must have been reached within 6 months of Step 2 registration. Resection extent will be recorded on the same basis described above for the low-risk group.
   * 1.1 In the setting of a newly diagnosed meningioma, the histologic diagnosis must have been reached within 24 weeks prior to Step 2 registration. In the setting of a recurrent meningioma, there are no such time constraints. Additional resection or biopsy is encouraged for patients with recurrence but is not requisite. If further biopsy or resection is performed at recurrence, these specimens must be submitted; submission of the original pathology specimens is encouraged but not required. The diagnosis of recurrence solely on the basis of imaging findings is permitted, but if no additional resection is performed, specimens from prior resection must be submitted.
   * 1.2 In cases of newly diagnosed or surgically treated recurrent meningioma, the operating neurosurgeon must provide a Simpson grade for the degree of resection.
2. History/physical examination, including neurologic examination, within 8 weeks prior to Step 2 registration
3. Zubrod Performance Status 0-1
4. Age ≥ 18
5. All patients must have a magnetic resonance imaging (MRI) scan within 12 weeks prior to Step 2 registration. Both preoperative and postoperative MRIs are required for all newly diagnosed patients in groups I, II, or III. In the setting of group II or III patients with recurrent/progressive meningioma and without recent surgery, a pre-operative study may not apply, although MRI documentation of recurrence or progression is required. MRIs must include precontrast T1, T2, and flair images and multiplanar (axial, sagittal, and coronal) postcontrast T1. The postoperative study must be completed within 12 weeks of surgery.

   * 5.1 Group I: All group I patients will have surgery. Preoperative and postoperative MRIs are thus required in order to assess resection extent.
   * 5.2 Group II: Surgery will be undertaken for the subgroup with a gross totally resected WHO grade II meningioma. For these patients preoperative and postoperative MRIs are necessitated. For the other subgroup with recurrent WHO grade I meningioma, preoperative and postoperative MRIs are required if surgery is undertaken for the recurrent/progressive tumor. However, only the follow-up imaging documenting recurrence or progression will apply if further surgery is not completed.
   * 5.3 Group III: Surgery will be undertaken for the subgroup with a newly diagnosed WHO grade III meningioma. For these patients preoperative and postoperative MRIs are obligatory. For the subgroups with recurrent WHO grade II or III meningioma, preoperative and postoperative MRIs are required if surgery is undertaken for the recurrent/progressive tumor. However, only the follow-up imaging documenting recurrence or progression will apply if further surgery is not completed.
6. For woman of childbearing potential who are intermediate or high risk:

   * 6.1 Negative serum pregnancy test within 14 days prior to Step 2 registration
   * 6.2 The patient must agree to practice adequate contraception from the time of the negative serum pregnancy test throughout the entire course of EBRT.
7. Patient must sign study-specific informed consent prior to study entry

Exclusion Criteria:

1. Extracranial meningioma
2. Multiple meningiomas
3. Hemangiopericytoma
4. Major medical illnesses or psychiatric impairments which, in the investigators opinion, will prevent administration or completion of the protocol therapy or preclude informed consent
5. Previous radiation therapy to the scalp, cranium, brain, or skull base
6. Prior invasive malignancy (except non-melanomatous skin cancer) unless disease free for a minimum of 3 years (for example, carcinoma in situ of the breast, oral cavity, or cervix are all permissible)
7. Patients with severe, active comorbidity including, but not restricted to:

   * 7.1 Unstable angina and/or congestive heart failure requiring hospitalization at the time of Step 2 registration
   * 7.2 Transmural myocardial infarction within the last 6 months
   * 7.3 Acute bacterial or fungal infection requiring intravenous antibiotics at the time of Step 2 registration
   * 7.4 Chronic obstructive pulmonary disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy at the time of Step 2 registration
   * 7.5 Hepatic insufficiency resulting in clinical jaundice and/or coagulation defects. Note, however, that laboratory tests for liver function and coagulation parameters are not required for entry into this protocol.
   * 7.6 Acquired immune deficiency syndrome (AIDS) based upon current Centers for Disease Control and Prevention (CDC) definition; note, however, that HIV testing is not required for entry into this protocol. The need to exclude patients with AIDS from this protocol is necessary because the treatments involved in this protocol may be significantly immunosuppressive.
   * 7.7 Active connective tissue disorders such as lupus or scleroderma if the patient is intermediate or high risk
8. Inability to receive gadolinium

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 244 (Actual)
Dates: Start 2009-06; Primary Completion 2016-09 (Actual); Study Completion 2023-08-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: C. Leland Rogers, MD, Principal Investigator — Virginia Commonwealth University
Locations (78):
- United States (74):
  - Arizona Oncology Services Foundation, Phoenix, Arizona
  - Mayo Clinic Hospital, Phoenix, Arizona
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Yale Cancer Center, New Haven, Connecticut
  - University of Florida Shands Cancer Center, Gainesville, Florida
  - Baptist-South Miami Regional Cancer Program, Miami, Florida
  - Emory Crawford Long Hospital, Atlanta, Georgia
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Curtis and Elizabeth Anderson Cancer Institute at Memorial Health University Medical Center, Savannah, Georgia
  - Saint Alphonsus Cancer Care Center at Saint Alphonsus Regional Medical Center, Boise, Idaho
  - Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois
  - Methodist Cancer Center at Methodist Hospital, Indianapolis, Indiana
  - Kansas Masonic Cancer Research Institute at the University of Kansas Medical Center, Kansas City, Kansas
  - Kansas City Cancer Centers - Southwest, Overland Park, Kansas
  - CCOP - Kansas City, Prairie Village, Kansas
  - Norton Suburban Hospital, Louisville, Kentucky
  - Mary Bird Perkins Cancer Center - Baton Rouge, Baton Rouge, Louisiana
  - Maine Center for Cancer Medicine and Blood Disorders - Scarborough, Scarborough, Maine
  - Greenebaum Cancer Center at University of Maryland Medical Center, Baltimore, Maryland
  - Baystate Regional Cancer Program at D'Amour Center for Cancer Care, Springfield, Massachusetts
  - Josephine Ford Cancer Center at Henry Ford Hospital, Detroit, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - St. Joseph Mercy Oakland, Pontiac, Michigan
  - Mercy Regional Cancer Center at Mercy Hospital, Port Huron, Michigan
  - Seton Cancer Institute at Saint Mary's - Saginaw, Saginaw, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Regions Hospital Cancer Care Center, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Kansas City Cancer Centers - South, Kansas City, Missouri
  - Kansas City Cancer Centers - North, Kansas City, Missouri
  - Siteman Cancer Center at Barnes-Jewish Hospital - Saint Louis, St Louis, Missouri
  - Billings Clinic - Downtown, Billings, Montana
  - Methodist Estabrook Cancer Center, Omaha, Nebraska
  - Nebraska Medical Center, Omaha, Nebraska
  - Norris Cotton Cancer Center at Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - CCOP - North Shore University Hospital, Manhasset, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - Highland Hospital of Rochester, Rochester, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - Albert Einstein Cancer Center at Albert Einstein College of Medicine, The Bronx, New York
  - Blumenthal Cancer Center at Carolinas Medical Center, Charlotte, North Carolina
  - Summa Center for Cancer Care at Akron City Hospital, Akron, Ohio
  - Barberton Citizens Hospital, Barberton, Ohio
  - Case Comprehensive Cancer Center, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Riverside Methodist Hospital Cancer Care, Columbus, Ohio
  - Grant Medical Center Cancer Care, Columbus, Ohio
  - Lake/University Ireland Cancer Center, Mentor, Ohio
  - Oklahoma University Cancer Institute, Oklahoma City, Oklahoma
  - Penn State Hershey Cancer Institute at Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Kimmel Cancer Center at Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Gibbs Regional Cancer Center at Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - University of Texas Medical Branch, Galveston, Texas
  - M. D. Anderson Cancer Center at University of Texas, Houston, Texas
  - Jon and Karen Huntsman Cancer Center at Intermountain Medical Center, Murray, Utah
  - Val and Ann Browning Cancer Center at McKay-Dee Hospital Center, Ogden, Utah
  - Huntsman Cancer Institute at University of Utah, Salt Lake City, Utah
  - Dixie Regional Medical Center - East Campus, St. George, Utah
  - Norris Cotton Cancer Center - North, Saint Johnsbury, Vermont
  - Virginia Commonwealth University Massey Cancer Center, Richmond, Virginia
  - University Cancer Center at University of Washington Medical Center, Seattle, Washington
  - St. Mary's Hospital Medical Center - Green Bay, Green Bay, Wisconsin
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Bay Area Cancer Care Center at Bay Area Medical Center, Marinette, Wisconsin
  - Community Memorial Hospital Cancer Care Center, Menomonee Falls, Wisconsin
  - Medical College of Wisconsin Cancer Center, Milwaukee, Wisconsin
  - Regional Cancer Center at Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Door County Cancer Center at Door County Memorial Hospital, Sturgeon Bay, Wisconsin
  - Waukesha Memorial Hospital Regional Cancer Center, Waukesha, Wisconsin
- Canada (4):
  - Cross Cancer Institute at University of Alberta, Edmonton, Alberta
  - Ottawa Hospital Regional Cancer Centre - General Campus, Ottawa, Ontario
  - Hopital Notre-Dame du CHUM, Montreal, Quebec
  - McGill Cancer Centre at McGill University, Montreal, Quebec

REFERENCES:
- [Result] Rogers CL, Perry A, Pugh S, Vogelbaum MA, Brachman D, McMillan W, Jenrette J, Barani I, Shrieve D, Sloan A, Bovi J, Kwok Y, Burri SH, Chao ST, Spalding AC, Anscher MS, Bloom B, Mehta M. Pathology concordance levels for meningioma classification and grading in NRG Oncology RTOG Trial 0539. Neuro Oncol. 2016 Apr;18(4):565-74. doi: 10.1093/neuonc/nov247. Epub 2015 Oct 22. PMID 26493095
- [Derived] Rogers CL, Won M, Vogelbaum MA, Perry A, Ashby LS, Modi JM, Alleman AM, Galvin J, Fogh SE, Youssef E, Deb N, Kwok Y, Robinson CG, Shu HK, Fisher BJ, Panet-Raymond V, McMillan WG, de Groot JF, Zhang P, Mehta MP. High-risk Meningioma: Initial Outcomes From NRG Oncology/RTOG 0539. Int J Radiat Oncol Biol Phys. 2020 Mar 15;106(4):790-799. doi: 10.1016/j.ijrobp.2019.11.028. Epub 2019 Nov 29. PMID 31786276
- [Derived] Rogers L, Zhang P, Vogelbaum MA, Perry A, Ashby LS, Modi JM, Alleman AM, Galvin J, Brachman D, Jenrette JM, De Groot J, Bovi JA, Werner-Wasik M, Knisely JPS, Mehta MP. Intermediate-risk meningioma: initial outcomes from NRG Oncology RTOG 0539. J Neurosurg. 2018 Jul;129(1):35-47. doi: 10.3171/2016.11.JNS161170. Epub 2017 Oct 6. PMID 28984517

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Two hundred forty-four patients registered for the first step registration which consisted of central pathology review confirmation of histology. One hundred seventy-eight continued on to the second step registration.
Groups:
- Intermidiate Risk: 54 Gy radiotherapy
Period: Overall Study
Arm/Group | Low Risk | Intermidiate Risk | High Risk
Started | 65 | 56 | 57
Completed | 60 | 52 | 53
Not Completed | 5 | 4 | 4
Not completed — Protocol Violation | 5 | 4 | 4

BASELINE CHARACTERISTICS:
Population: All eligible patients
Groups:
- Total: Total of all reporting groups
Arm/Group | Low Risk | Intermidiate Risk | High Risk | Total
Number analyzed (Participants) | 60 | 52 | 53 | 165
Age, Continuous [Median (Full Range); unit: years] | 56 [31 to 79] | 53 [18 to 73] | 62 [19 to 94] | 56 [18 to 94]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 32 | 28 | 108
  Male | 12 | 20 | 25 | 57

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival Rate at 3 Years
Description: Progression was determined by central review of magnetic resonance imaging (MRI) exams and is defined as an increase in measurable tumor of greater than 20% in any diameter, or as new nodular enhancement in patients with no measurable tumor on initial postoperative imaging. In the absence of neurologic progression (NP), suspected imaging progression of less than 5 mm (maximum diameter) must be confirmed on two successive follow-up MRI studies, a minimum of 3 months apart. NP is defined as a new or progressive neurologic deficit attributed to the meningioma, with or without measurable meningioma growth. Progression-free survival (PFS) rates are estimated using the binomial method.
Time Frame: From registration to 3 years
Population: Eligible patients who started study treatment and evaluable for 3-year progression-free survival
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Low Risk | Intermidiate Risk | High Risk
Number analyzed (Participants) | 51 | 48 | 51
percentage of participants | 92.2 [81.1 to 97.8] | 93.7 [82.8 to 98.7] | 58.8 [44.2 to 72.4]

2. Secondary Outcome: Number of Patients With Grades 2-5 Acute Adverse Events in the Following Categories Individually and Combined: Neurology, Ocular/Visual, Dermatologic/Skin [Excluding Alopecia]
Description: Grades 2-5 neurology, ocular/visual, dermatologic/skin [excluding alopecia] categories, individually and combined for acute adverse events as assessed by NCI Common Toxicity Criteria for Adverse Effects (CTCAE) v3.0 where the attribution is related to treatment as definite, probable, possible, or unknown. Adverse events are graded using CTCAE v3.0. Grade refers to the severity of the AE. The CTCAE v3.0 assigns Grades 1 through 5 with unique clinical descriptions of severity for each AE based on this general guideline: Grade 1 Mild AE, Grade 2 Moderate AE, Grade 3 Severe AE, Grade 4 Life-threatening or disabling AE, Grade 5 Death related to AE.
Time Frame: From start of radiation to 90 days.
Population: Eligible patients who started study treatment with acute AE assessed. Low risk patients are not reported since they did not receive any study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Intermidiate Risk | High Risk
Number analyzed (Participants) | 46 | 53
Participants
  Neurology: Grade 2 | 4 | 3
  Neurology: Grade 3 | 0 | 2
  Neurology: Grade 4 | 0 | 0
  Neurology: Grade 5 | 0 | 0
  Neurology: None Grade 2-5 | 42 | 48
  Ocular/visual: Grade 2 | 1 | 0
  Ocular/visual: Grade 3 | 0 | 0
  Ocular/visual: Grade 4 | 0 | 0
  Ocular/visual: Grade 5 | 0 | 0
  Ocular/visual: None Grade 2-5 | 45 | 53
  Dermatology/Skin: Grade 2 | 1 | 2
  Dermatology/Skin: Grade 3 | 0 | 0
  Dermatology/Skin: Grade 4 | 0 | 0
  Dermatology/Skin: Grade 5 | 0 | 0
  Dermatology/Skin: None Grade 2-5 | 45 | 51
  Groups combined: Grade 2 | 5 | 4
  Groups combined: Grade 3 | 0 | 2
  Groups combined: Grade 4 | 0 | 0
  Groups combined: Grade 5 | 0 | 0
  Groups combined: None Grade 2-5 | 41 | 47

3. Secondary Outcome: Number of Patients With Grades 2-5 Late Adverse Events in the Following Categories Individually and Combined: Neurology, Ocular/Visual, Dermatologic/Skin [Excluding Alopecia]
Description: Grades 2-5 neurology, ocular/visual, dermatologic/skin [excluding alopecia] categories, individually and combined for acute adverse events as assessed by NCI Common Toxicity Criteria for Adverse Effects (CTCAE) v3.0 where the attribution is related to treatment as definite, probable, possible, or unknown. Late adverse events are those occurring more than 90 days from start of radiation therapy.
Time Frame: Ninety-one days from start of radiation therapy to last follow-up. Maximum follow-up at time of analysis was 6.3 years.
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Intermidiate Risk | High Risk
Number analyzed (Participants) | 51 | 51
Participants
  Neurology: Grade 2 | 12 | 11
  Neurology: Grade 3 | 0 | 3
  Neurology: Grade 4 | 0 | 0
  Neurology: Grade 5 | 0 | 1
  Neurology: None Grade 2-5 | 39 | 36
  Ocular/visual: Grade 2 | 0 | 0
  Ocular/visual: Grade 3 | 0 | 0
  Ocular/visual: Grade 4 | 0 | 0
  Ocular/visual: Grade 5 | 0 | 0
  Ocular/visual: None Grade 2-5 | 51 | 51
  Dermatology/Skin: Grade 2 | 1 | 0
  Dermatology/Skin: Grade 3 | 0 | 0
  Dermatology/Skin: Grade 4 | 0 | 0
  Dermatology/Skin: Grade 5 | 0 | 0
  Dermatology/Skin: None Grade 2-5 | 50 | 51
  Groups combined: Grade 2 | 13 | 11
  Groups combined: Grade 3 | 0 | 3
  Groups combined: Grade 4 | 0 | 0
  Groups combined: Grade 5 | 0 | 1
  Groups combined: None Grade 2-5 | 38 | 36

4. Secondary Outcome: Overall Survival Rate at 3 Years
Description: Overall survival time is defined as time from randomization to date of death from any cause and is estimated by the Kaplan-Meier method. Patients last known to be alive are censored at the date of last contact.
Time Frame: From registration to 3 years
Population: Eligible patients who started study treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Low Risk | Intermidiate Risk | High Risk
Number analyzed (Participants) | 52 | 48 | 51
percentage of participants | 98.1 [89.7 to 100.0] | 95.8 [85.8 to 99.5] | 78.4 [64.7 to 88.7]

5. Secondary Outcome: Progression-free Survival Rate at 3 Years (Kaplan-Meier Method)
Description: Progression was determined by central review of MRI exams and is defined as an increase in measurable tumor of greater than 20% in any diameter, or as new nodular enhancement in patients with no measurable tumor on initial postoperative imaging. In the absence of neurologic progression (NP), suspected imaging progression of less than 5 mm (maximum diameter) must be confirmed on two successive follow-up MRI studies, a minimum of 3 months apart. NP is defined as a new or progressive neurologic deficit attributed to the meningioma, with or without measurable meningioma growth. Progression-free survival time is defined as time from registration to the date of progression, death, or last known follow-up (censored). Progression-free survival rates are estimated using the Kaplan-Meier method.
Time Frame: From registration to 3 years
Population: Eligible patients who started study treatment and evaluable for 3-year progression-free survival
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Low Risk | Intermidiate Risk | High Risk
Number analyzed (Participants) | 60 | 52 | 53
percentage of participants | 91.4 [84.2 to 98.6] | 93.9 [87.2 to 100.0] | 59.2 [45.7 to 72.6]

6. Secondary Outcome: Number of Participants Determined to Have MRI Imaging Features as Assessed by Central Neuroradiology Review at Diagnosis, at Progression, and at 3 Years
Description: MRI's were centrally reviewed by the study neuroradiology co-chairs for presence of edema, homogeneous enhancement, calcification, hyperostosis, and brain invasion. Data is presented for all risk groups combined, with time points presented in each column. Neither risk groups nor time points are compared.
Time Frame: Baseline, at time of first progression, and at 3 years
Population: Eligible participants who started study treatment, had a centrally reviewed MRI at the given time, and whose MRI was evaluable for the given feature
Measure: Count of Participants; unit: Participants
Arm/Group | MRI at Diagnosis | MRI at First Progression | MRI at 3 Years
Number analyzed (Participants) | 148 | 23 | 79
Participants
  Edema: number analyzed (Participants) | 114 | 18 | 39
  Edema | 76 | 13 | 15
  Homogeneous Enhancement: number analyzed (Participants) | 116 | 12 | 33
  Homogeneous Enhancement | 88 | 9 | 14
  Calcification: number analyzed (Participants) | 27 | 5 | 20
  Calcification | 6 | 0 | 1
  Hyperostosis: number analyzed (Participants) | 40 | 5 | 20
  Hyperostosis | 17 | 0 | 1
  Brain Invasion: number analyzed (Participants) | 30 | 8 | 22
  Brain Invasion | 1 | 0 | 1

7. Secondary Outcome: Greatest Single Dimension From MRI as Assessed by Central Neuroradiology Review at Diagnosis, at Progression, and at 3 Years
Description: MRI's were centrally reviewed by the study neuroradiology co-chairs. Data is presented for all risk groups combined, with time points presented in each column. Neither risk groups nor time points are compared.
Time Frame: Baseline, at time of first progression, and at 3 years
Population: Eligible participants who started study treatment, had a centrally reviewed MRI at the given time, and whose MRI was evaluable for tumor dimension.
Measure: Median (Full Range); unit: milimeters
Arm/Group | MRI at Diagnosis | MRI at First Progression | MRI at 3 Years
Number analyzed (Participants) | 148 | 21 | 28
milimeters | 42.7 [4.2 to 144.4] | 34.7 [14.0 to 104.0] | 29.0 [7.5 to 129.9]

8. Secondary Outcome: Adherence to Protocol-specific Target and Normal Tissue Radiotherapy Parameters
Description: The principle investigator performed a radiotherapy quality assurance (QA) review.
Time Frame: After treatment delivery
Population: Eligible participants who started treatment and were centrally reviewed
Measure: Count of Participants; unit: Participants
Arm/Group | Intermidiate Risk | High Risk
Number analyzed (Participants) | 44 | 46
Participants
  Per protocol | 36 | 39
  Acceptable variation | 4 | 5
  Unacceptable deviation | 2 | 1
  Not evaluable | 2 | 1

9. Secondary Outcome: Concordance Between Central and Parent Institution Histopathologic Grading/Subtyping
Description: A pathology review was conducted both by the institution and centrally, with three possible choices for grade / subtype: World Health Organization (WHO) Grade I / benign; WHO grade II / atypical; WHO grade III / anaplastic. Data is presented for all risk groups combined.
Time Frame: Baseline
Population: Eligible patients with central and site reviews
Measure: Count of Participants; unit: Participants
Arm/Group | Central Review: Benign | Central Review: Atypical | Central Review: Anaplastic
Number analyzed (Participants) | 76 | 71 | 25
Participants
  Site Review: Benign | 74 | 9 | 1
  Site Review: Atypical | 2 | 60 | 8
  Site Review: Anaplastic | 0 | 2 | 16
Statistical Analysis 1: Comparison: Central Review: Benign vs Central Review: Atypical vs Central Review: Anaplastic; The Kappa (κ) coefficient was used to assess the measure of agreement between the reviewers. κ can be interpreted as follows (κ / Agreement): < 0 / Less than chance agreement; 0.01-0.20 / Slight agreement; 0.21-0.40 / Fair agreement; 0.41-0.60 / Moderate agreement; 0.61-0.80 / Substantial agreement; 0.81-0.99 / Almost perfect agreement. The asymptotic test of the null hypothesis: κ=0 will be performed using the Z-statistic to determine the strength of agreement; Test type: Other; p < 0.0001, Z test; Kappa statistic = 0.79, 95% CI 2-sided [0.71 to 0.87]

10. Secondary Outcome: Molecular Correlative Studies
Time Frame: From registration to 3 years
Population: The protocol did not provide sufficient detail to meet National Cancer Institute requirements for release of specimens from the NRG Oncology tissue bank for the protocol-specified analysis, therefore no assays were performed and no data were collected for this outcome measure. Specimen use will require federal approval and funding separate from this trial.
Arm/Group | Intermidiate Risk | High Risk
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Histopathologic Correlates of PFS Including Light Microscopy, Immunohistochemical Analysis, and Microarray Analysis
Time Frame: From registration to 3 years
Population: The protocol did not provide sufficient detail to meet National Cancer Institute requirements for release of specimens from the NRG tissue bank for the protocol-specified analysis, therefore no assays were performed and no data were collected for this outcome measure. Specimen use will require federal approval and funding separate from this trial.
Arm/Group | Intermidiate Risk | High Risk
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: Eligible patients who started protocol treatment. Subjects experiencing more than one of a given adverse event are counted only once for that adverse event.
Arm/Group | Low Risk | Intermidiate Risk | High Risk
All-Cause Mortality (participants affected / at risk) | 22/60 | 47/52 | 47/53
Serious Adverse Events (participants affected / at risk) | 0/60 | 1/52 | 5/53
Other Adverse Events (participants affected / at risk) | 22/60 | 47/52 | 47/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Low Risk (N=60) | Intermidiate Risk (N=52) | High Risk (N=53)
Gait abnormal (General disorders) | 0 | 0 | 1
Pain [other] (General disorders) | 0 | 0 | 1
Soft tissue infection [with normal or Grade 1-2 ANC] (Infections and infestations) | 0 | 0 | 1
Central nervous system necrosis (Nervous system disorders) | 0 | 1 | 1
Neurological disorder NOS (Nervous system disorders) | 0 | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 1
Seizure (Nervous system disorders) | 0 | 0 | 2
Tremor (Nervous system disorders) | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Low Risk (N=60) | Intermidiate Risk (N=52) | High Risk (N=53)
Hemoglobin decreased (Blood and lymphatic system disorders) | 0 | 1 | 6
Hearing loss (Ear and labyrinth disorders) | 0 | 8 | 4
Tinnitus (Ear and labyrinth disorders) | 0 | 4 | 0
Eye disorder (Eye disorders) | 1 | 5 | 3
Flashing vision (Eye disorders) | 0 | 3 | 1
Vision blurred (Eye disorders) | 2 | 7 | 6
Constipation (Gastrointestinal disorders) | 0 | 4 | 5
Diarrhea (Gastrointestinal disorders) | 0 | 4 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 3 | 2
Nausea (Gastrointestinal disorders) | 0 | 11 | 11
Vomiting (Gastrointestinal disorders) | 0 | 5 | 1
Edema limbs (General disorders) | 0 | 0 | 4
Fatigue (General disorders) | 5 | 34 | 29
Gait abnormal (General disorders) | 0 | 1 | 5
General symptom (General disorders) | 0 | 3 | 0
Dermatitis radiation (Injury, poisoning and procedural complications) | 0 | 6 | 9
Radiation recall reaction (dermatologic) (Injury, poisoning and procedural complications) | 0 | 2 | 8
Lymphocyte count decreased (Investigations) | 0 | 0 | 4
Platelet count decreased (Investigations) | 1 | 1 | 4
Weight loss (Investigations) | 0 | 5 | 2
Anorexia (Metabolism and nutrition disorders) | 0 | 7 | 6
Blood glucose increased (Metabolism and nutrition disorders) | 1 | 0 | 7
Serum albumin decreased (Metabolism and nutrition disorders) | 0 | 0 | 4
Serum calcium decreased (Metabolism and nutrition disorders) | 0 | 0 | 4
Serum potassium decreased (Metabolism and nutrition disorders) | 1 | 0 | 4
Serum sodium decreased (Metabolism and nutrition disorders) | 0 | 0 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 4 | 3
Muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 5
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 3 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 4 | 2
Ataxia (Nervous system disorders) | 1 | 3 | 3
Central nervous system necrosis (Nervous system disorders) | 0 | 0 | 3
Cognitive disturbance (Nervous system disorders) | 1 | 3 | 7
Dizziness (Nervous system disorders) | 5 | 14 | 9
Headache (Nervous system disorders) | 10 | 25 | 21
Memory impairment (Nervous system disorders) | 4 | 8 | 14
Neurological disorder NOS (Nervous system disorders) | 1 | 1 | 7
Olfactory nerve disorder (Nervous system disorders) | 0 | 3 | 0
Peripheral motor neuropathy (Nervous system disorders) | 1 | 3 | 3
Peripheral sensory neuropathy (Nervous system disorders) | 5 | 6 | 7
Seizure (Nervous system disorders) | 4 | 7 | 14
Speech disorder (Nervous system disorders) | 2 | 3 | 8
Taste alteration (Nervous system disorders) | 0 | 3 | 6
Tremor (Nervous system disorders) | 0 | 1 | 3
Anxiety (Psychiatric disorders) | 3 | 2 | 3
Depression (Psychiatric disorders) | 4 | 4 | 8
Insomnia (Psychiatric disorders) | 2 | 4 | 2
Urinary frequency (Renal and urinary disorders) | 0 | 3 | 2
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 6
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 28 | 32
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 2 | 5
Rash desquamating (Skin and subcutaneous tissue disorders) | 0 | 0 | 3
Scalp pain (Skin and subcutaneous tissue disorders) | 3 | 0 | 3
Skin disorder (Skin and subcutaneous tissue disorders) | 0 | 2 | 3
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 4 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI's are required to abide by the sponsor's publication guidelines which require review by coauthors and subsequent review and approval by the sponsor.